CLINICAL TRIAL: NCT01940939
Title: Study of Repetitive Transcranial Magnetic Stimulation in the Treatment of Cognitive Impairment in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11ZR1431600
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Active Comparator): Active treatment will be delivered at an intensity that is 90% of the resting motor threshold (RMT). Stimulation will be delivered at 20 Hz with 100 stimulation trains of 20 stimuli each (i.e., 2000 stimuli) and an inter-train interval of 9 sec. Treatment will be applied in sequential order to the left dorsolateral prefrontal cortex (DLPFC). Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but the coil will be reversed. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The MagPro X100 is connected to a Magnetic Coil which transfers the magnetic stimulation to the tissue. The original coils MC-B65 can be used with the MagPro X100.

SUMMARY:
1. Exploration of repetitive transcranial magnetic stimulation（rTMS）on working memory and cognitive impairment symptoms of schizophrenia treatment and mechanism.
2. Analysis of high-frequency repetitive transcranial magnetic stimulation stimulation to the improvement of negative symptoms and psychotic symptoms.

DETAILED DESCRIPTION:
The study was a randomized double-blind sham-controlled trial for 4 weeks. Patients with schizophrenia were treated with 20-Hz rTMS for 4 weeks to the left dorsolateral prefrontal cortex (added to the ongoing treatment). Negative symptoms were assessed with the Scale for the Assessment of Negative Symptoms (SANS), the Positive and Negative symptom scale (PANSS).The auditory steady state responses (ASSR) were obtained for the assessment of gamma oscillation.And cognitive symptoms were assessed by MATRICS cognitive test battery (MCCB) Chinese version and n-back task.

ELIGIBILITY:
Inclusion Criteria:

* 1）patients to be diagnosed according to the Fourth Edition of the Diagnostic and Statistical Manual of Mental Disorders(DSM-IV) for paranoid schizophrenia；2）20～49 years old；3）Duration of 2 ~ 10 years;4）the disease situation is stable， the fluctuation of Positive and Negative Symptom Scale（PANSS）total score ≤10% in last 1 month, and have accepted the current drugs for more than 8 weeks; 5）Patients, their families and doctors are agreed that the disease situation is stable and maintained current drug treatment in next month；6）Signed an informed consent

Exclusion Criteria:

* 1)patients to be diagnosed according to DSM-IV for substance abused,development delayed;2)suffering from serious physical disease and can not accept the treatment;3)repetitive transcranial magnetic stimulation(rTMS) contraindications: intracranial metal substance, with heart pacemakers and cochlear implants, intracranial pressure;4)the disease situation is not stable， the fluctuation of Positive and Negative Symptom Scale（PANSS）total score >10% in last 1 month, Positive and Negative Symptom Scale（PANSS）total score > 60;5)difficult to maintain the current drug treatment for at least 1 month;6）undergoing electroconvulsive therapy（ECT）in last 3 months.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dengtang Liu, MD, Study Director — Chief Psychiatrist and Professor
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhuo K, Tang Y, Song Z, Wang Y, Wang J, Qian Z, Li H, Xiang Q, Chen T, Yang Z, Xu Y, Fan X, Wang J, Liu D. Repetitive transcranial magnetic stimulation as an adjunctive treatment for negative symptoms and cognitive impairment in patients with schizophrenia: a randomized, double-blind, sham-controlled trial. Neuropsychiatr Dis Treat. 2019 May 8;15:1141-1150. doi: 10.2147/NDT.S196086. eCollection 2019. PMID 31190822

RESULTS

PARTICIPANT FLOW:
Groups:
- Active rTMS: Active treatment will be delivered at an intensity that is 80% of the resting motor threshold (RMT). Stimulation will be delivered at 20 Hz with 100 stimulation trains of 20 stimuli each (i.e., 2000 stimuli) and an inter-train interval of 9 sec. Treatment will be applied in sequential order to the left dorsolateral prefrontal cortex (DLPFC). Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Repetitive Transcranial Magnetic Stimulation: The MagPro X100 is connected to a Magnetic Coil which transfers the magnetic stimulation to the tissue. The original coils MC-B65 can be used with the MagPro X100.
- Sham rTMS: Sham rTMS stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but the coil will be reversed. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Repetitive Transcranial Magnetic Stimulation: The MagPro X100 is connected to a Magnetic Coil which transfers the magnetic stimulation to the tissue. The original coils MC-B65 can be used with the MagPro X100.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 35 | 35
Completed | 33 | 27
Not Completed | 2 | 8
Not completed — Withdrawal by Subject | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 22 | 25 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Severity of Negative Symptoms
Description: The assessment of negative symptoms were measured with the Positive and Negative Symptom Scale (PANSS) and the Scale for the Assessment of Negative Symptoms (SANS).The SANS contains 30 particular items divided into 5 symptomatological domains: 1) affective flattening and/or blunting, 2) alogia, 3) avolition and/or apathy, 4) anhedonia, and 5) impaired attention. Each item is scored on a scale from 0 (not at all) to 5 (severe) with a total scoring range of 0 to 150. Higher scores indicate more impairment.The PANSS contains 30 particular items divided into 3 subscores: 1)positive, 2) negative, and 3) general subscore. Each item is scored on a scale from 1 (absent) to 7 (extreme) with a total scoring range of 30 to 210. Higher scores indicate more impairment. The primary outcomes were the changes in the severity of negative symptoms as measured with SANS total score and PANSS negative subscore after 4 weeks of intervention.
Time Frame: Baseline, after 4 weeks of treatment
Population: Ten patients dropped out due to different reasons (three patients refused to participated, three did not complianted and the other four were discharged before completion of study)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 33 | 27
units on a scale
  SANS（Baseline） | 48.09 [31 to 78] | 50.33 [35 to 91]
  SANS（4 weeks） | 33.91 [23 to 54] | 41.00 [24 to 70]
  PANSS（Baseline） | 68.15 [60 to 82] | 69.93 [61 to 82]
  PANSS（4 weeks） | 54.58 [40 to 73] | 59.85 [48 to 76]

2. Secondary Outcome: MATRICS Consensus Cognitive Battery (MCCB) in Chinese Version
Description: MCCB in Chinese Version includes 9 tasks across 7 domains, and a composite score, including Processing Speed (Brief Assessment of Cognition in Schizophrenia Symbol Coding, Animal Fluency, Trails A), Attention (Continuous Performance Test), Working Memory (WMS-III Spatial Span), Verbal Learning (Hopkins Verbal Learning Test - Revised), Visual Learning (Brief Visuospatial Memory Test - Revised), Problem Solving (Neuropsychological Assessment Battery), and Social Cognition (Mayer-Salovey- Caruso Emotional Intelligence Test).The results are reported as T scores with a mean of 50 and an SD of 10.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MCCB(T score)
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 33 | 27
MCCB(T score)
  Composite score (baseline) | 45.07 (6.48) | 43.58 (9.25)
  Composite score (4 weeks) | 48.00 (7.16) | 49.04 (7.46)

3. Other Pre Specified Outcome: Event-related Spectral Perturbation (ERSP)
Description: Alterations in gamma-band ASSR have been thought to be the most robust finding of abnormal neural oscillations in patients with schizophrenia. EEG data were acquired using a 64-electrode cap and alternating current BrainAmp amplifiers (Brain Products GmbH, Germany). We used EEGLAB to perform time-frequency analysis with a short-term Fourier transformation, and then calculated ERSP.
Time Frame: 4 weeks
Population: patients discontinualed treatment
Measure: Mean (Full Range); unit: dB
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 14
dB
  baseline | 0.365 [0.079 to 0.706] | 0.327 [0.046 to 0.669]
  4 weeks | 0.390 [0.251 to 0.721] | 0.382 [0.052 to 0.711]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Sham rTMS: 3 subjects reported a transient headache in the initial period, After giving comfort the symptoms were significantly reduced.
  No other adverse events were observed.
- Active rTMS: 4 subjects reported a transient headache and 1 subjects reported dizziness in the initial period.After giving comfort and reducing initial intensity of stimulation, the symptoms were significantly reduced.
  No other adverse events were observed.
Arm/Group | Sham rTMS | Active rTMS
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 3/35 | 5/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham rTMS (N=35) | Active rTMS (N=35)
headache (General disorders) | 3 (3) | 4 (4)
dizzsiness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No